CLINICAL TRIAL: NCT02960854
Title: Randomized, Double-Blind, Parallel Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-936558 (Nivolumab) in Participants With Severe Sepsis or Septic Shock.
Brief Title: A Study of Nivolumab Safety and Pharmacokinetics in Patients With Severe Sepsis or Septic Shock.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CA209-923
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nivolumab 1 (Experimental): Dose 1
  Interventions: Biological: Nivolumab
- Nivolumab 2 (Experimental): Dose 2
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558

SUMMARY:
A study to evaluate the safety, tolerability and pharmacokinetics of Nivolumab in participants with severe sepsis or septic shock.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women ages ≥ 18 years old
* Documented or suspected infection
* Severe sepsis or septic shock for at least 24 hours
* Sepsis-induced immunosuppression
* In Intensive Care Unit (ICU) with no plans to discharge in next 24 hours

Exclusion Criteria:

* Previous episode of severe sepsis or septic shock with ICU admission during the current hospitalization
* Autoimmune disease
* Organ or bone marrow transplant
* Cancer treatment in the past 6 weeks
* Human immunodeficiency virus (HIV) infection and not on therapy prior to this episode of sepsis; hepatitis C virus(HCV) infection and still has virus (not cured); Chronic hepatitis B virus (HBV) infection and not on treatment

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (16):
  - Uc Davis Medical Center, Sacramento, California
  - Univ. Of Colorado Health, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - University Of Florida, Gainesville, Florida
  - Pulmonary And Critical Care Of Atlanta, Atlanta, Georgia
  - Osf Saint Francis Medical Center, Peoria, Illinois
  - University Of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Division of Acute Care Surgery, Ann Arbor, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Hotchkiss RS, Colston E, Yende S, Crouser ED, Martin GS, Albertson T, Bartz RR, Brakenridge SC, Delano MJ, Park PK, Donnino MW, Tidswell M, Mayr FB, Angus DC, Coopersmith CM, Moldawer LL, Catlett IM, Girgis IG, Ye J, Grasela DM. Immune checkpoint inhibition in sepsis: a Phase 1b randomized study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of nivolumab. Intensive Care Med. 2019 Oct;45(10):1360-1371. doi: 10.1007/s00134-019-05704-z. Epub 2019 Oct 1. PMID 31576433
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 subjects were enrolled in the study. 31 were randomized; 7 not randomized: (5) Failed to meet study eligibility criteria, (1) died, (1) withdrew consent
Groups:
- Nivolumab (480 mg): the assessment of the safety and tolerability of a single dose of nivolumab 480 mg
- Nivolumab (960 mg): the assessment of the safety and tolerability of a single dose of nivolumab 960 mg
Period: Overall Study
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Started | 15 | 16
Completed | 8 | 7
Not Completed | 7 | 9
Not completed — Not Disclosed | 2 | 2
Not completed — Subject No Longer Meets Study Criteria | 1 | 0
Not completed — Subject Withdrew Consent | 0 | 1
Not completed — Death | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg) | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (12.30) | 58.4 (15.16) | 57.5 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Incidence Rates of Serious Adverse Events (SAEs), Adverse Events (AEs), Immune-mediated AEs, AEs Leading to Discontinuation, and Deaths
Time Frame: Screening, day -1, day 1 and subsequent days after, up to 90 days
Population: All treated participants
Measure: Number; unit: Percentage
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
Percentage
  Serious Adverse Events (SAEs) | 6.7 | 43.8
  Adverse Events (AEs) | 93.3 | 87.5
  Immune-Mediated Adverse Events | 53.3 | 81.3
  AEs leading to discontinuation | 0.0 | 0.0
  Deaths | 40.0 | 38.7

2. Primary Outcome: Composite of Vital Signs and Electrocardiogram (ECG)
Description: Includes body temperature, respiratory rate, blood pressure and heart rate. Blood pressure and heart rate should be measured after the participant has been resting quietly for at least 5 minutes.
Time Frame: Screening up to 90 days (Discharge)
Population: All treated participants
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
Percentage
  ECG Change from Baseline (Discharge) | -18.0 (31.68) | -29.0 (3.46)
  Vital Signs - Diastolic Pressure (mmHg) Screening | 61.5 (20.37) | 58.5 (9.00)
  Vital Signs - Systolic Pressure (mmHg) Screening | 116.5 (21.48) | 105.5 (14.65)
  Vital Signs - Heart Rate (beats/min) Screening | 80.1 (21.34) | 94.6 (16.64)
  Vital Signs - Resp. Rate (breaths/min) Screening | 23.0 (6.08) | 24.4 (8.83)
  Vital Signs - Temperature (C) Screening | 37.19 (0.79) | 37.11 (0.77)
  Vital Signs - Diastolic Pressure (mmHg) Discharge: number analyzed (Participants) | 6 | 4
  Vital Signs - Diastolic Pressure (mmHg) Discharge | 79.7 (16.49) | 70.5 (16.28)
  Vital Signs - Systolic Pressure (mmHg) Discharge: number analyzed (Participants) | 6 | 4
  Vital Signs - Systolic Pressure (mmHg) Discharge | 129.0 (25.06) | 110.0 (16.47)
  Vital Signs - Heart Rate (beats/min) Discharge: number analyzed (Participants) | 6 | 4
  Vital Signs - Heart Rate (beats/min) Discharge | 85.3 (18.89) | 86.5 (19.76)
  Vital Signs - Resp. Rate (breaths/min) Discharge: number analyzed (Participants) | 6 | 4
  Vital Signs - Resp. Rate (breaths/min) Discharge | 18.8 (2.71) | 17.5 (3.32)
  Vital Signs - Temperature (C) Discharge: number analyzed (Participants) | 6 | 4
  Vital Signs - Temperature (C) Discharge | 36.60 (0.276) | 36.90 (0.337)

3. Primary Outcome: Peak Nivolumab Serum Concentration (Cmax)
Description: Participants peak nivolumab serum concentration
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All Treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
ug/mL | 123 (85.4) | 246 (85.4)

4. Primary Outcome: Trough Nivolumab Serum Concentration (Cmin)
Description: Participant trough nivolumab serum concentration
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
ug/mL | 21.6 (39) | 43.2 (39)

5. Primary Outcome: Average Nivolumab Serum Concentration (Cavg)
Description: Participant average nivolumab serum concentration
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
ug/mL | 42.7 (28.5) | 85.4 (28.5)

6. Primary Outcome: Time of Maximum Observed Concentration (Tmax)
Description: Participant observed time of maximum concentration
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All Treated participants
Measure: Median (Full Range); unit: hours
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
hours | 1.67 [1.47 to 24.3] | 1.53 [1.37 to 48.0]

7. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration [AUC(0-T)]
Description: Area under the serum concentration-time curve from time zero to time of last quantifiable concentration
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
h*ug/mL | 18099 (51) | 32130 (83)

8. Primary Outcome: Total Clearance (CLT)
Description: Total clearance of serum concentration of nivolumab
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
L/h | 0.025 (50) | 0.027 (85)

9. Primary Outcome: Volume of Distribution (Vd)
Description: Vlume of distribution of nivolumab serum concentration
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
L | 12.0 (42) | 13.3 (54)

10. Primary Outcome: Half-life (T1/2)
Description: Half-Life of nivolumab derived from serum concentration
Time Frame: Day 1 and subsequent days after, up to 90 days
Population: All Treated Participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
hours | 353 (126.5) | 378 (189.6)

11. Secondary Outcome: Receptor Occupancy
Description: Receptor occupancy on T cells at baseline and after study treatment administration at planned sampling time points
Time Frame: Day 1 and up to day 90 (discharge)
Population: All Treated Participants
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
Percentage
  Baseline: number analyzed (Participants) | 13 | 16
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Study Discharge: number analyzed (Participants) | 7 | 4
  Study Discharge | 81.272 (27.69) | 71.14 (34.83)

12. Secondary Outcome: Number of Participants With Detectable Anti-nivolumab Antibodies
Description: Participant with positive anti-drug antibody detection
Time Frame: Baseline and subsequent days after, up to 90 days
Population: All Treated Participants
Measure: Number; unit: Percentage
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
Percentage | 73.3 | 75.0

13. Secondary Outcome: Number of Participants With Any Detectable Anti-drug Antibodies
Time Frame: Baseline and subsequent days after, up to 90 days
Population: All Treated Participants
Measure: Number; unit: Percentage
Arm/Group | Nivolumab (480 mg) | Nivolumab (960 mg)
Number analyzed (Participants) | 15 | 16
Percentage | 26.7 | 56.3

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from Day 1 following single dose of nivolumab, up until Day 90.
Groups:
- NIVOLUMAB 480mg: the assessment of the safety and tolerability of a single dose of nivolumab 480 mg
- NIVOLUMAB 960mg: the assessment of the safety and tolerability of a single dose of nivolumab 960 mg
Arm/Group | NIVOLUMAB 480mg | NIVOLUMAB 960mg
All-Cause Mortality (participants affected / at risk) | 4/15 | 6/16
Serious Adverse Events (participants affected / at risk) | 1/15 | 7/16
Other Adverse Events (participants affected / at risk) | 14/15 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 480mg (N=15) | NIVOLUMAB 960mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Electrocardiogram st segment elevation (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 480mg (N=15) | NIVOLUMAB 960mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 6 | 8
Bandaemia (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 4
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 2
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiomegaly (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Mastoid effusion (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Corneal epithelium defect (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Pupils unequal (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Asthenia (General disorders) | 1 | 0
Catheter site haematoma (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Generalised oedema (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 2
Pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 6
Secretion discharge (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Porcelain gallbladder (Hepatobiliary disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 1
Candida infection (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Genital infection fungal (Infections and infestations) | 1 | 0
Herpes dermatitis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Purulent discharge (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Viral tracheitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Stoma site discharge (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Ammonia increased (Investigations) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase abnormal (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2
Bacterial test positive (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood bilirubin abnormal (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 1
Breath sounds abnormal (Investigations) | 1 | 1
Bronchoalveolar lavage abnormal (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Chest x-ray abnormal (Investigations) | 1 | 1
Clostridium test positive (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram qt prolonged (Investigations) | 1 | 1
Fungal test positive (Investigations) | 0 | 1
Gastric ph increased (Investigations) | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Herpes simplex test positive (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 2
Lipase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1
Oxygen saturation decreased (Investigations) | 2 | 1
Reticulocyte count increased (Investigations) | 0 | 1
Sputum culture positive (Investigations) | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 2
White blood cell count increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 3
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 4
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Thrombosis in device (Product Issues) | 1 | 0
Agitation (Psychiatric disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Dry gangrene (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 6 | 4
Labile blood pressure (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02960854/SAP_000.pdf
  • Study Protocol (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02960854/Prot_001.pdf